CLINICAL TRIAL: NCT01046474
Title: Preventing Excessive Weight Gain by Reducing Carbonated Beverage and Sugar Consumption and Increasing Physical Activity Among Public School Adolescents From the Metropolitan Area of Rio de Janeiro
Brief Title: Reducing Beverages and Sugar and Increasing Physical Activity in Public School Adolescents From Brazil
Acronym: PAPAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Rosely Sichieri, State University of Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMS-PAPAS-project
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Sugar Intake; Beverage Intake; Fruit Intake; Beans Intake; Physical Activity
Keywords: school children; body mass index; sugar intake; beverage intake
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- reducing beverages and sugar and increase physical activity (Experimental): reduction of beverages and sugar and increasing physical activity
  Interventions: Behavioral: lifestyle
- control -no intervention (No Intervention)

INTERVENTIONS:
Behavioral: lifestyle — Based on beliefs and behaviors of children sections of education will be delivered via classroom activities.
  Activities will be facilitated by trained research assistants. Printed instructions and orientations on the facilitation process will support the assistants' efforts. The activities will require 20 to 30 minutes, and teachers will be encouraged to reiterate the message during their lesson. The goal is to promote ten one-hour sessions of activity for each class.
  Children will also be stimulated to increase everyday activities such as walking and playing games at home and school. Also, activities with parents and family members such as walking around the neighborhood on weekends will be promoted.
  Arms: reducing beverages and sugar and increase physical activity

SUMMARY:
The main objective is to evaluate the effect on BMI of a school-based program that discourages the consumption of all sweetened beverages, encourages the reduction in sugar intake, and encourages the increase in physical activity among adolescents and their families from a low socioeconomic area.

DETAILED DESCRIPTION:
Specific objectives are:

1. To compare total, lean, and fatty body mass variation in adolescents aged 11 to 14, from 7th and 8th grades from schools under intervention and from the ones not subjected to the intervention program.
2. To compare sweetened beverages consumption and sugar intake before and after the intervention in both groups of schools.
3. To evaluate the impact of the intervention on the selling of sweetened beverages in the cafeterias.
4. To compare change in family expenditures with sweetened beverages and sugar.

ELIGIBILITY:
Inclusion Criteria:

* 5th grades

Exclusion Criteria:

* Pregnancy

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Body mass index | one year

SECONDARY OUTCOMES:
Mean lean and fatty body mass proportions: measured by portable electrical bioimpedance bean | one year

CONTACTS AND LOCATIONS:
Locations (1):
- 20 Schools of Metropolitan Area, Duque de Caxias, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Munoz-Espinosa LE, Torre A, Cisneros L, Montalvo I, Male R, Mejia S, Aguilar JR, Lizardi J, Zuniga-Noriega J, Eugenia Icaza M, Gasca-Diaz F, Hernandez-Hernandez L, Cordero-Perez P, Chi L, Torres L, Rodriguez-Alvarez F, Tapia G, Poo JL. Noninvasive Evaluation of Prolonged-Release Pirfenidone in Compensated Liver Cirrhosis. ODISEA Study, a Randomised Trial. Liver Int. 2025 Jun;45(6):e70131. doi: 10.1111/liv.70131. PMID 40402087
- [Derived] Cunha DB, de Souza Bda S, Pereira RA, Sichieri R. Effectiveness of a randomized school-based intervention involving families and teachers to prevent excessive weight gain among adolescents in Brazil. PLoS One. 2013;8(2):e57498. doi: 10.1371/journal.pone.0057498. Epub 2013 Feb 25. PMID 23451237